CLINICAL TRIAL: NCT03090685
Title: Effects of Auriculotherapy on Pain and Functional Capacity of Individuals With Chikungunya Fever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Bernardo Diniz Coutinho, Department of Physical Therapy, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1193-8428
Record Dates: First submitted 2017-03-14; First posted 2017-03-27 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Chikungunya Fever
Keywords: Chikungunya Fever; Pain; Mobility Limitation; Auriculotherapy; Complementary Therapies; Physical Therapy
MeSH Terms: conditions — Chikungunya Fever; Pain; Mobility Limitation | interventions — Seeds

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind randomized controlled trial (RCT).
Who Masked: Participant, Outcomes Assessor
Masking Description: The sample randomization procedure will be performed by means of a computer program, which will generate a random sequence to be placed in an opaque envelope by an assistant not involved in the evaluation and treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True auriculotherapy with seeds (Experimental): Auriculotherapy complementary to the usual drug treatment. At each ear, selected points edible seeds of roasted mustard with a size of approximately 2 mm will be used, since it is natural and non-toxic. The seeds will be stored in ear plate and applied with the use of micropore clamp and tape in 4 to 5 specific points to control for musculoskeletal pain.
  Interventions: Procedure: True auriculotherapy with seeds
- Placebo Auriculotherapy with seeds (Placebo Comparator): Placebo Auriculotherapy complementary to usual drug treatment. Seeds will be used in 4 auricular points in the lobe of the ear that have no specific relation to the musculoskeletal pain in the lower limbs and with the innervation of the vagus nerve.
  Interventions: Procedure: Placebo Auriculotherapy with seeds

INTERVENTIONS:
Procedure: True auriculotherapy with seeds — Roasted edible mustard seeds with ~ 2mm diameter fixed with adhesive tape in 4 to 5 specific body points to control musculoskeletal pain.
  Other Names: Auriculotherapy complementary to the drug therapy
  Arms: True auriculotherapy with seeds
Procedure: Placebo Auriculotherapy with seeds — Roasted edible mustard seeds with ~ 2mm diameter fixed with adhesive tape at 4 points located in the auricular lobe not specific for musculoskeletal pain.
  Other Names: Placebo Auriculotherapy complementary to usual treatment
  Arms: Placebo Auriculotherapy with seeds

SUMMARY:
Chikungunya fever is an acute viral disease, transmitted by the mosquito (Aedes aegypti), that triggers pain and disabling rheumatic manifestations. There is no cure for this disease, and the usual treatment is directed at relieving symptoms through the use of analgesics and antipyretics. Due to the risk of adverse effects triggered by prolonged use of analgesic and anti-inflammatory drugs, the use of complementary therapies, such as Auriculotherapy, might be a safe and effective non-pharmacological treatment for the management of Chikungunya symptomatic cases.

Subjects diagnosed with Chikungunya and undergoing routine treatment will receive auricotherapy treatment once a week, for five weeks. Subjects will be assessed at baseline and after 4 and 8 weeks after intervention. This study might help understand the use of Auriculotherapy as a complementary treatment in the treatment of physical and functional symptoms of individuals infected by Chikungunya .

DETAILED DESCRIPTION:
Objectives of the study

1. To evaluate the effectiveness of Auriculotherapy in the management of pain and functional capacity of symptomatic individuals after Chikungunya fever.
2. To evaluate the effects of Auriculotherapy on the intensity of pain, limitation of mobility, and perception of disability and physical capacity.
3. Investigate the effect of Auriculotherapy on pain medication use.

Place and study population: Subjects diagnosed with Chikungunya Fever will be recruited for convenience in the basic care of the city of Fortaleza-CE, Brazil, in order to be evaluated and treated by the researcher's team.

Procedures and intervention: Subjects will be evaluated at the initial time of the research, and after 4 and 8 weeks of intervention. The description of the procedures will follow the guidelines of the Consolidated Standards of Reporting Trials (CONSORT) and the Standards for Reporting Interventions in Controlled Trials of Acupuncture (STRICTA). Asepsis of the ear with alcohol 70%is necessary to apply 4 to 5 auricular acupuncture points. In the intervention group, specific points will be used to the management of pain and physical function. In the placebo group, non-specific points will be used. Patients will be instructed to exert finger pressure at each point for 3 minutes. At least 3x / day, or whenever they feel pain. These implants will be kept for 5 days and will be taken off by the participant 2 days before the next appointment.

Ethical aspects: The research will begin after approval by the Ethics and Research Committee (CEP) of the Federal University of Ceará. All participants will sign the Informed Consent and are free to withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged ≥ 18 years;
* with medical or other referral from the Family Health Strategy due to symptoms resulting from Chikungunya fever confirmed by clinical or laboratory criteria;
* be able to understand instructions and answer the questions asked by the interviewer.

Exclusion Criteria:

* complaints of pain unrelated to the lower limbs;
* presence of malignant neoplastic disease;
* history of traumatic injury or the lower limb and surgery in the last 12 months;
* congenital deformation;
* pregnancy;
* history of treatment with with Auriculotherapy, acupuncture or physiotherapy in the last four weeks;
* use of steroid medication in the last month;
* use of opioids during the study period;
* do not sign the Free and Informed Consent Form (TCLE).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Pain Numerical rating scale (NRS) | collected at baseline up to 2 months after therapy
  Graded scale from 0 (no pain) to 10 (worst pain imaginable) that evaluates in one-dimensional the perception of pain by asking about the average pain felt in the past seven days in the symptomatic limb.
Timed Up and Go Test (TUG) | collected at baseline up to 2 months after therapy
  Performance-based test designed to assess functional mobility and risk of falls in frail older adults.This instrument has been associated with other to test musculoskeletal conditions.

SECONDARY OUTCOMES:
World Health Disability Assessment Schedule (WHODAS 2.0) | collected at baseline up to 2 months after therapy
  Generic instrument with high internal consistency (α: 0.86), high test-retest reliability (ICC: 0.98) that evaluates deficiency and functionality based on six domains (cognition, mobility, self-care, interpersonal relations, life activity and participation).
Short Physical Performance Battery (SPPB) | collected at baseline up to 2 months after therapy
  Test consisted of thress sub-tests that assess the functional capacity of the lower limbs, through static balance, gait speed and lower limb muscle strength.
Reducing the use of pain medication | collected at baseline up to 2 months after therapy
  Patient self-report on the use of analgesic and anti-inflammatory drugs, by recording the dosage and type of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Renata N Kirkwood, doctor, Study Director — Federal University of Minas Gerais
Locations (1):
- Grupo de Atenção Integral e Pesquisa em Acupuntura e Medicina Tradicional Chinesa - GAIPA, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No